CLINICAL TRIAL: NCT07256509
Title: A Phase II Study to Evaluate the Safety and Efficacy of SYS6010 Combined With Osimertinib Versus Osimertinib as Neoadjuvant Therapy in Participants With Resectable Stage II-IIIB Non-squamous Non-small Cell Lung Cancer With EGFR Mutation Positive
Brief Title: A Study of SYS6010 Combined With Osimertinib Versus Osimertinib Alone as Neoadjuvant Therapy for Patients With EGFR Mutation-positive Resectable Non-squamous Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS6010-013
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Randomized, Open-label, Phase II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYS6010 + Osimertinib (Experimental): Neoadjuvant Therapy: SYS6010 + Osimertinib Adjuvant Therapy: Osimertinib + Pemetrexed + Cisplatin or Carboplatin
  Interventions: Drug: SYS6010; Drug: Osimertinib
- Osimertinib (Active Comparator): Neoadjuvant Therapy: Osimertinib Adjuvant Therapy: Osimertinib + Pemetrexed + Cisplatin or Carboplatin
  Interventions: Drug: Osimertinib; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: SYS6010 — SYS6010 by intravenous (IV) infusion
  Arms: SYS6010 + Osimertinib
Drug: Osimertinib — Osimertinib, oral
  Other Names: Osimertinib Mesylate Tablets
Drug: Pemetrexed — 500 mg/m^2 by IV infusion, Q3W
  Arms: Osimertinib
Drug: Cisplatin — 75 mg/m^2 by IV infusion, Q3W
  Arms: Osimertinib
Drug: Carboplatin — AUC 5 mg/mL•min by IV infusion, Q3W
  Arms: Osimertinib

SUMMARY:
To evaluate the safety and efficacy of SYS6010 combined with osimertinib as neoadjuvant therapy for patients with resectable EGFR mutation non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
This study includes three stages: a neoadjuvant therapy stage, a surgery stage, and an adjuvant follow-up stage. In the neoadjuvant therapy stage, eligible participants will be stratified by stage (Stage II and Stage III) and mutation type (19Del and L858R) and randomized in a 1:1 ratio to the SYS6010 combined with osimertinib treatment group and the osimertinib monotherapy group. Neoadjuvant therapy will be administered for 3 cycles.

In the surgery stage, the feasibility of surgery will be assessed by a thoracic surgery investigator. Surgery should be performed between Week 10 and Week 12 (i.e., D64-D84 after the first dose of neoadjuvant therapy). Tumor samples collected during surgery will be sent to a central pathology laboratory to assess pathological response.

In the adjuvant therapy stage, all participants who undergo surgery will subsequently enter the adjuvant therapy stage. Participants who do not undergo surgery for reasons other than disease progression will also enter the adjuvant therapy stage.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign the written informed consent form (ICF);
2. Age 18-75 years, regardless of sex;
3. Histologically or cytologically confirmed non-squamous non-small cell lung cancer, staged as resectable or potentially resectable Stage II-IIIB disease according to the International Association for the Study of Lung Cancer (IASLC) 8th Edition TNM staging criteria;
4. Must be eligible for complete surgical resection of the primary tumor;
5. Nodal status must be evaluated by whole-body FDG-PET and contrast-enhanced CT;
6. Confirmed presence of an EGFR-sensitizing mutation (exon 19 deletion or exon 21 L858R mutation, co-mutation with other EGFR sites is allowed), as tested by a central laboratory or local testing facility;
7. No prior systemic anti-tumor therapy (including chemotherapy, biotherapy, targeted therapy, immunotherapy);
8. At least one measurable lesion at baseline as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
9. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
10. Life expectancy ≥6 months;
11. Adequate major organ and bone marrow function;
12. Women or men of childbearing potential must use highly effective contraception.

1. Able to understand and voluntarily sign the written informed consent form (ICF); 2. Age 18-75 years, regardless of sex; 3. Histologically or cytologically confirmed non-squamous non-small cell lung cancer, staged as resectable or potentially resectable Stage II-IIIB disease according to the International Association for the Study of Lung Cancer (IASLC) 8th Edition TNM staging criteria; 4. Must be eligible for complete surgical resection of the primary tumor; 5. Nodal status must be evaluated by whole-body FDG-PET and contrast-enhanced CT; 6. Confirmed presence of an EGFR-sensitizing mutation (exon 19 deletion or exon 21 L858R mutation, co-mutation with other EGFR sites is allowed), as tested by a central laboratory or local testing facility; 7. No prior systemic anti-tumor therapy (including chemotherapy, biotherapy, targeted therapy, immunotherapy); 8. At least one measurable lesion at baseline as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1; 9. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1; 10. Life expectancy ≥6 months; 11. Adequate major organ and bone marrow function; 12. Women or men of childbearing potential must use highly effective contraception.

Exclusion Criteria:

1. Diagnosis of Stage I, Stage IIIB with N3, and Stage IIIC, IVA, and IVB non-small cell lung cancer;
2. Multiple primary malignancies (refer to exclusion criterion #8 for synchronous primary lung cancer) OR a mixed histology of SCLC and NSCLC;
3. T4 stage lung cancer due to invasion of the great vessels, carina, trachea, esophagus, heart, or vertebral body; and/or bulky N2 disease;
4. Eligible only for segmentectomy or wedge resection;
5. Receipt of Chinese patent medicine preparations indicated for the treatment of lung cancer within 1 week before randomization;
6. Major surgery or severe traumatic injury within 4 weeks before the first study treatment, or expected to undergo major surgery during the study period;
7. History of other primary malignant tumor (including any known or suspected concurrent primary lung cancer);
8. History of autoimmune disease, immunodeficiency, or organ transplant (except for corneal transplant);
9. Refractory nausea, vomiting, chronic gastrointestinal disease, inability to swallow drugs orally;
10. Evidence of severe or uncontrolled medical conditions (including uncontrolled hypertension, diabetes mellitus, etc,);
11. Active or prior history of interstitial lung disease (ILD)/pneumonitis;
12. Expected to receive live vaccine therapy within 30 days after randomization;
13. History of a definite neurological or mental disorder; known allergy, hypersensitivity, or intolerance to the study drugs or any of their excipients;
14. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) Rate | Within 8 weeks post-surgery
  Defined as the proportion of participants with ≤10% residual viable tumor cells in the resected primary tumor bed, as assessed by blinded independent pathological review (BIPR).
Pathological Complete Response (pCR) Rate | Within 8 weeks post-surgery
  The proportion of participants with no residual viable tumor cells in both the resected primary tumor bed and lymph nodes, as assessed by BIPR.
Downstaging from N2 to N0/N1 or N1 to N0 at the time of surgery | Within 8 weeks post-surgery
Disease-Free Survival (DFS) | Up to approximately 5.5 years after the last participant enrolled
  Investigator-assessed DFS per RECIST v1.1
Event-Free Survival (EFS) | Up to approximately 5.5 years after the last participant enrolled
  Investigator-assessed DFS per RECIST v1.1
Objective Response Rate (ORR) | Up to approximately 5.5 years after the last participant enrolled
  Investigator-assessed ORR per RECIST v1.1
Overall Survival (OS) | Up to approximately 5.5 years after the last participant enrolled
Incidence of Adverse Events (AEs) | Up to approximately 5.5 years after the last participant enrolled
Anti-drug Antibodies (ADAs) to SYS6010 | Up to approximately 5.5 years after the last participant enrolled